CLINICAL TRIAL: NCT05512546
Title: Coil Embolization and Thromboembolic Complications in Patients With Ruptured Aneurysms
Brief Title: The Prevention of Thromboembolic Complications Associated With Coil Embolization
Status: Completed | Type: Observational
Sponsor: Muhammad Hassan (Other)
Responsible Party: Sponsor-Investigator, Muhammad Hassan, Registrar Neurology, Shaheed Zulfiqar Ali Bhutto Medical University
Organization: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Other Study IDs: Lahore General Hospital
Record Dates: First submitted 2022-08-21; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Thromboembolic Stroke; Aspirin; Clopidogrel; Coil Embolization; Prevention
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Aspirin Group: patients were prescribed 75 mg/day of either aspirin for 6 months
  Interventions: Drug: Aspir-Low Pill
- Clopidogrel Group: 75mg/day prescribed for 6 months
  Interventions: Drug: Aspir-Low Pill

INTERVENTIONS:
Drug: Aspir-Low Pill — patients were prescribed 75 mg/day of either aspirin

SUMMARY:
Clopidogrel has been to be reported to be superior to aspirin for the prevention of thromboembolic complications associated with coil embolization in patients with ruptured aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* All the patients enrolled in the study underwent MRI and Angiography.
* Participants included in the study were confirmed on assessment, and verified for ruptured aneurysm by imaging using either computed tomography (CT) or MRI.

Exclusion Criteria:

* Patients with any history of sensitivity or reaction to aspirin, or any contraindication for MRI, were excluded from the study.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with ruptured cerebral hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
High Intensity Areas | at 24 hours
  post procedural
High Intensity Areas | 3 months
  Post Procedural

SECONDARY OUTCOMES:
High Intensity Areas | at 6 months
  Post procedural

CONTACTS AND LOCATIONS:
Overall Officials: Umair Rasheed, FRCPS, Study Director — Lahore General Hospital
Locations (1):
- Umair Rasheed, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided